CLINICAL TRIAL: NCT03220529
Title: A Study to Test the Potential of Brillouin Microscopy for Biomechanical Properties Measurements in Human Cornea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Seok Hyun Yun, Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P002404
Record Dates: First submitted 2017-06-09; First posted 2017-07-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Pellucid Marginal Corneal Degeneration; Keratoconus; Keratectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Normal healthy subjects (Active Comparator): Healthy subjects with normal appearing corneas respecting all the general inclusion/exclusion criteria. Multiple axial measurements with the Brillouin Ocular Scanner on the cornea will be carried out.
  Interventions: Device: Brillouin Ocular Scanner
- Keratoconus subjects (Active Comparator): Subjects classified as patients with mild, moderate, or advanced keratoconus. Multiple axial measurements with the Brillouin Ocular Scanner on the cornea will be carried out.
  Interventions: Device: Brillouin Ocular Scanner
- Subjects diagnosed with PMD (Active Comparator): Subjects with Pellucid marginal corneal degeneration (PMD). Multiple axial measurements with the Brillouin Ocular Scanner on the cornea will be carried out.
  Interventions: Device: Brillouin Ocular Scanner
- Patients before and after LASK surgery (Active Comparator): Healthy subjects who are scheduled to undergo LASIK surgery. Multiple axial measurements with the Brillouin Ocular Scanner on the cornea will be carried out.
  Interventions: Device: Brillouin Ocular Scanner
- Patients with keratoconus before and after CXL (Active Comparator): Subjects who are scheduled to undergo collagen crosslinking treatment. Multiple axial measurements with the Brillouin Ocular Scanner on the cornea will be carried out.
  Interventions: Device: Brillouin Ocular Scanner

INTERVENTIONS:
Device: Brillouin Ocular Scanner

SUMMARY:
The purpose of this research study is to find out if the new Brillouin Ocular Scanner can measure the variation (difference) of the corneal elastic changes involved in the onset of corneal ectasia, induced by LASIK surgery and cornea collagen crosslinking (CXL) treatment. Ectasia refers to the thinning and bulging of the cornea and results in severe vision degradation (loss), which may occur because of a progressive disease (keratoconus) or because of LASIK surgery. It is believed that the structural weakening of the cornea plays a major role in developing ectasia. CXL is a treatment that is able to halt the progression of ectasia.

The Brillouin Ocular Scanner is a technique based on the principles used in the laser speed measuring of a car (radar gun). When laser light illuminates a moving sample, a portion of the light slightly changes color. In our body, e.g in eye and corneal tissue, very weak sound waves are naturally present and they can induce a similar color shift. Measuring this color shift with a sensitive light color meter (spectrometer), we will measure the sound speed in the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with healthy cornea
* Patients with mild, moderate, or advanced keratoconus
* Subjects diagnosed with PMD
* Patients before and after LASK surgery
* Patients with keratoconus before and after collagen crosslinking treatment

Exclusion Criteria:

* Normal volunteer group: presbyopia and/or cataract
* Keratoconus subjects group: corneas with scars developed, received any ocular surgery, such as laser vision correction surgeries or CXL treatment
* Subjects diagnosed with PMD: excludes corneas received any ocular surgery, such as laser vision correction or CXL treatment
* Patients before and after LASK surgery Corneas received priori ocular surgeries, taking any ocular medications except season allergy medicine such as artificial tears

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Brillouin frequency shift of corneal stroma | at time of measurement
  Brillouin frequency shift of corneal stroma in normal corneas and corneas diagnosed with keratoconus and pellucid marginal degeneration
Change of Brillouin frequency shift from base line in corneas received LASIK surgery | 1 day and 4-8 weeks
  Brillouin frequency shift in corneas before and after receiving LASIK surgery
Change of Brillouin frequency shift from base line in corneas received crosslinking treatment | 3 days, 1 month, 3 months, 6 months
  Brillouin frequency shift in corneas before and after receiving crosslinking surgery

CONTACTS AND LOCATIONS:
Overall Officials: Seok Hyun Yun, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States
- Institute for Refractive and Ophthalmic Surgery, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scarcelli G, Besner S, Pineda R, Kalout P, Yun SH. In vivo biomechanical mapping of normal and keratoconus corneas. JAMA Ophthalmol. 2015 Apr;133(4):480-2. doi: 10.1001/jamaophthalmol.2014.5641. No abstract available. PMID 25611213
- [Background] Scarcelli G, Besner S, Pineda R, Yun SH. Biomechanical characterization of keratoconus corneas ex vivo with Brillouin microscopy. Invest Ophthalmol Vis Sci. 2014 Jun 17;55(7):4490-5. doi: 10.1167/iovs.14-14450. PMID 24938517
- [Background] Scarcelli G, Pineda R, Yun SH. Brillouin optical microscopy for corneal biomechanics. Invest Ophthalmol Vis Sci. 2012 Jan 20;53(1):185-90. doi: 10.1167/iovs.11-8281. PMID 22159012
- [Background] Scarcelli G, Polacheck WJ, Nia HT, Patel K, Grodzinsky AJ, Kamm RD, Yun SH. Noncontact three-dimensional mapping of intracellular hydromechanical properties by Brillouin microscopy. Nat Methods. 2015 Dec;12(12):1132-4. doi: 10.1038/nmeth.3616. Epub 2015 Oct 5. PMID 26436482